CLINICAL TRIAL: NCT02769273
Title: Stellarex Vascular E-Registry
Acronym: SAVER
Status: Completed | Type: Observational
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: D029260
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: RCC 2-3
  Interventions: Device: Percutaneous Transluminal Angioplasty
- Cohort 2: RCC 4-6 (CLI)
  Interventions: Device: Percutaneous Transluminal Angioplasty

INTERVENTIONS:
Device: Percutaneous Transluminal Angioplasty
  Other Names: Stellarex™ OTW Drug-coated Angioplasty Balloon

SUMMARY:
Prospective, international, multi-center, single arm, observational study to continue to assess the treatment by the Stellarex™ OTW Drug-coated Angioplasty Balloon in superficial femoral and/or popliteal arteries according to the Instructions for Use in a broad, real-world, claudicant or ischemic rest pain patients population per the institution's standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients intended to be treated with Stellarex for de-novo or restenotic lesions of the femoro-popliteal arteries
* Rutherford Clinical Category (RCC) 2-3 or 4 indicated for a Percutaneous Transluminal Angioplasty according to local applicable guidelines
* Patients intended to be treated with Stellarex for de-novo or restenotic lesions of the superficial femoral, popliteal and/or infra-popliteal arteries*
* Rutherford Clinical Category (RCC) 2-6 indicated for a Percutaneous Transluminal Angioplasty according to local applicable guidelines
* Age ≥18 years old
* Life expectancy > 1 year
* Is able and willing to provide written informed consent prior to enrollment in the study (as applicable)
* Is able and willing to come on site or to be contacted by phone for the follow-up

Exclusion Criteria:

Patients with any medical condition that would make him/her inappropriate for treatment with Stellarex as per Instructions for Use (IFU) or investigator's opinion

* Patient already enrolled in other investigational (interventional) studies that would interfere with study endpoints
* Patients with severe disease of foot circulation defined as:

  * "desert foot" (absence of any angiographically visible arterial network below the ankle)
  * Or lack of a patent (<50%DS) and hemodynamically relevant wound related arterial pathway in the foot
* Patients confined to bed that are completely non ambulatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic stenosis of the superficial femoral artery and/or popliteal artery intended to be treated with a Percutaneous Transluminal Angioplasty using the Stellarex OTW Drug -Coated Balloon
Sampling Method: Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2016-06; Primary Completion 2021-10-31 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint Cohort 1 - RCC 2-3: | 12 months post-procedure
  Freedom from clinically-driven Target Lesion Revascularization (CD-TLR) at 12 months post- procedure.
Primary Safety Endpoint-Cohort 1 - RCC 2-3 | 30 days post-procedure - 12Month post procedure
  Freedom from device and procedure- related death through 30 days post-procedure and freedom from target limb major amputation and CD-TLR through 12 months post-procedure.
Primary effectiveness endpoint: Cohort 2 - RCC 4-6 (CLI) | 6 Months post procedure
  Freedom from CD-TLR at 6 months post-procedure.
Primary safety endpoint-Cohort 2 - RCC 4-6 (CLI) | 30days
  Freedom from Composite MALE and POD through 30 days

SECONDARY OUTCOMES:
Rate and Freedom from events as specified in the description :Cohort 1 - RCC 2-3 | as specified in the description
  * All-cause mortality at 12, 24 and 36 months post- procedure
  * Cardiovascular death at 12, 24, 36 months post- procedure
  * Procedural complication defined as occurrence of death, stroke, myocardial infraction, emergent surgical revascularization, significant distal embolization in target limb, or thrombosis of target vessel through the end of the procedure
  * Device or procedure related death at 30 days
  * Major target limb amputation at 12, 24, 36 months post-procedure
  * CD-TLR through 12 (rate only), 24 and 36 months
  * Clinically Driven- Target Vessel Revascularization (CD- TVR) through 12, 24 and 36 months
Rate and Freedom-from-Cohort 2 - RCC 4-6 | As specified in the description
  All-cause mortality at 6, 12, 24 and 36 months post- procedure
  * Cardiovascular death at 6, 12, 24, 36 months post- procedure
  * Procedural complication defined as occurrence of death, stroke, myocardial infraction, emergent surgical revascularization, significant distal embolization in target limb, or thrombosis of target vessel through the end of the procedure
  * Device or procedure related death at 30 days o Major target limb amputation at 6, 12, 24, 36 months post-procedure
  * CD-TLR through 6 (rate only), 12, 24 and 36 months o Clinically Driven- Target Vessel Revascularization (CD- TVR) through 6, 12, 24 and 36 months
  * Wound healing rate through 6, 12, 24, and 36 months post-procedure
  * Minor amputation through 6, 12, 24 and 36 months
  * Amputation-free survival through 6, 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Locations (46):
- Austria (3):
  - Medical University Graz, Graz
  - Krankenhaus der Barmherzigen Schwesterrn Reid, Ried im Innkreis
  - Krankenhaus Göttlicher Heiland GmbH, Vienna
- Belgium (9):
  - UZA Antwerpen, Edegem, Edegem
  - OLV Aalst, Aalst
  - Imelda, Bonheiden
  - Europe Hospital, Brussels
  - AZ Sint Blasius, Dendermonde
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis Hasselt, Hasselt
  - AZ Groeninge, Kortrijk
  - H.Hart Tienen, Tienen
- France (10):
  - Clinique Générale Annecy, Annecy
  - Clinique Rhone Durance, Avignon
  - Clinique Saint Augustin, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Clinique Médipole De Savoie, Challes-les-Eaux
  - Grand Hôpital de l'Est Francilien - Site de Marne la Vallée, Jossigny
  - Groupe hospitalier Saint Joseph, Paris
  - Polyclinique de la Baie, Saint-Martin-des-Champs
  - Clinique Pasteur, Toulouse
  - Clinique Sarrus teinturiers Rive Gauche, Toulouse
- Germany (13):
  - Klinikum Arnsberg, Arnsberg
  - Ev. Krankenhaus Königin Elisabeth Herzberge, Berlin
  - MediClin Herzzentrum Coswig, Coswig
  - Klinikum Doebeln GmbH, Döbeln
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Krankenhäuser Landkreis Freudenstadt GmbH, Freudenstadt
  - Universitätsklinikum Halle, Halle
  - Asklepios Klinikum Harburg, Hamburg
  - Universitätsklinikum Jena, Jena
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Universitätsklinikum Leipzig, Leipzig
  - Saint Vincenz Hospital, Limburg
  - St. Franziskus-Hospital GmbH, Münster
- Italy (6):
  - Âzienda Ospedaliera Per L'emergenza Cannizzaro, Catania
  - AZ Ospedaliera M. Mellini Chiari, Chiari
  - Clinica Montevergine, Mercogliano
  - Ospedale Civile Di Mirano, Mirano
  - Multimedica, Sesto San Giovanni
  - "Villa Berica" Gruppo Garofalo, Vicenza
- United Kingdom (5):
  - The Royal Bournemouth Hospital, Bournemouth
  - North Bristol NHS Trust, Bristol
  - Stoke Mandeville Hospital, Buckingham
  - "Saint George's Vascular Institute, London
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024